CLINICAL TRIAL: NCT03349346
Title: Phase 1b Trial Evaluating Idelalisib in Children and Adolescents With Relapsed or Refractory Diffuse Large B-cell Lymphoma or Mediastinal B-cell Lymphoma in Combination With RICE
Brief Title: Idelalisib With Rituximab, Ifosfamide, Carboplatin, Etoposide (RICE) in Children and Adolescents
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The European Medical Agency granted a Paediatric Investigational Product-specific waiver on the grounds that idelalisib is likely to be unsafe in paediatrics
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-313-1090; 2017-001468-39 (EudraCT Number)
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diffuse Large B-Cell Lymphoma; Mediastinal B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — idelalisib; Rituximab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1- Participants 12 to less than 18 years of age (Experimental): Participants will receive idelalisib monotherapy (from day 1 to day 21), followed by combination therapy with RICE. Upon enrollment, participants will be assigned to one of the 3 dose levels during idelalisib monotherapy (Dose level 1 = 55 mg/m^2 twice daily (BID), Dose level 2 = 85 mg/m^2 BID, Dose level 3 = 125 mg/m^2 BID) administered as 50 mg, 100 mg or 150 mg tablets as appropriate, or as 10 mg dispersible tablets for oral suspension for participants who cannot swallow tablets.
  * Day 1: single dose of idelalisib
  * Day 2 up to Day 21: initiate and continue idelalisib BID dosing
  * Day 22 for up to 12 months: idelalisib twice per day in combination with RICE. Cycles of RICE will be administered over 5 days every 3 weeks (Day 1: rituximab; Day 3: rituximab, ifosfamide, carboplatin, etoposide; Days 4 and 5: ifosfamide, etoposide) starting day 22 (or earlier if there is evidence of clinical progression while on idelalisib monotherapy) for up to 12 months.
  Interventions: Drug: Idelalisib; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide
- Cohort 2- Participants 1 to less than 12 years of age (Experimental): Participants will receive one of the 3 doses of idelalisib monotherapy (from day 1 to day 21) followed by combination therapy with RICE. Idelalisib will be administered as as 50 mg, 100 mg or 150 mg tablets as appropriate, or as 10 mg dispersible tablets for oral suspension for participants who cannot swallow tablets. Participants will will be enrolled at dose level 1 once tolerability is demonstrated in the older cohort (Cohort 1). Thereafter, both age cohorts will be dose escalated independently.
  * Day 1: single dose of idelalisib
  * Day 2 up to Day 21: initiate and continue idelalisib BID
  * Day 22 for up to 12 months: idelalisib twice per day in combination with RICE. Cycles of RICE will be administered over 5 days every 3 weeks (Day 1: rituximab; Day 3: rituximab, ifosfamide, carboplatin, etoposide; Days 4 and 5: ifosfamide, etoposide) starting day 22 (or earlier if there is evidence of clinical progression while on idelalisib monotherapy) for up to 12 months.
  Interventions: Drug: Idelalisib; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Idelalisib — Tablet (s) or dispersible tablets for suspension administered orally twice daily
  Other Names: Zydelig®
Drug: Rituximab — 375 mg/m^2 administered intravenously
Drug: Ifosfamide — 3 mg/m^2 administered intravenously
Drug: Carboplatin — 635 mg/m^2 administered intravenously
Drug: Etoposide — 100 mg/m^2 administered intravenously

SUMMARY:
The primary objectives of this study are to evaluate safety, tolerability, pharmacokinetics (PK) and preliminary efficacy of idelalisib; and to establish recommended phase 2 doses (RP2D) of idelalisib in combination with rituximab, ifosfamide, carboplatin, etoposide (RICE) in children and adolescents with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) or mediastinal B-cell lymphoma (MBCL)

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of DLBCL or MBCL established by the World Health Organization (WHO) 2008 classification of tumors of hematopoietic and lymphoid tissues
* Relapsed or refractory disease
* Measurable or evaluable disease based on imaging or bone marrow examination
* Karnofsky ≥ 60% for participants > 16 years of age or Lansky ≥ 60 for participants ≤ 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* A negative serum pregnancy test is required for females of child bearing potential.
* Participants of child bearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception .
* Lactating females must agree to discontinue nursing before idelalisib is administered
* Adequate bone marrow function as defined in the protocol
* Adequate renal function as defined in the protocol

Key Exclusion Criteria:

* Prior ifosfamide, carboplatin, etoposide (ICE) therapy, with or without an anti-CD20 antibody, or history of hypersensitivity to any components of RICE
* Known active central nervous system or leptomeningeal lymphoma or within 4 weeks from the last intrathecal therapy prior to the required diagnostic lumbar puncture (LP) for this study
* Disease progression within 6 months from last anti-CD20 therapy
* Ongoing toxicity from prior cytotoxic therapy (last dose at least 3 weeks prior to study entry)
* Less than 4 half-lives from the last dose of previous targeted therapy and ongoing acute toxicity of prior targeted therapy
* Active infection with human immunodeficiency virus (HIV), cytomegalovirus (CMV), hepatitis B virus (HBV), or hepatitis C virus (HCV) based on screening serology and polymerase chain reaction (PCR) results
* Evidence of systemic bacterial, fungal, or viral infection at the time of treatment start (Day 1)
* Ongoing or history of drug-induced pneumonitis
* Ongoing or history of inflammatory bowel disease
* Pregnancy or breastfeeding
* Currently receiving other anti-cancer or other investigational drug
* Prior solid organ transplantation
* Prior allogeneic stem cell transplantation within 60 days or active acute graft versus host disease (GVHD) Grade 3 or higher
* Known hypersensitivity to idelalisib, the metabolites, or formulation excipients
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with the study requirements

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of Dose Limiting Toxicities (DLTs) | Up to Day 21
  DLTs refer to toxicities experienced during the first 21 days of study treatment that have been judged to be clinically significant and related to study treatment.
Proportion of Participants Experiencing Adverse Events (AEs) | Up to 12 months
Proportion of Participants Experiencing Serious Adverse Events (SAEs) | Up to 12 months
Proportion of Participants Experiencing Adverse Events (AEs) Leading to Idelalisib Interruption, Idelalisib Dose Reduction, Premature Discontinuation of Idelalisib, or Death | Up to 12 months

SECONDARY OUTCOMES:
Rate of Grade ≥ 3 Transaminase Elevations Based on Laboratory Findings | Up to 12 months
Overall Response Rate (ORR) | Up to 12 months
  Overall response rate (ORR) is defined as the proportion of participants who achieve a best response of Complete Response (CR) or Partial Response (PR) after the first dose of idelalisib (either as a result of monotherapy or in combination with RICE chemoimmunotherapy). The screening imaging study will serve as the reference for ORR.
Overall Survival (OS) | Up to 5 years
  Overall Survival (OS) is defined as the interval from the first dose date of idelalisib to death from any cause.
Progression-Free Survival (PFS) | Up to 12 months
  Progression-Free Survival (PFS) is defined as the interval from the start date of RICE to the earlier of the first documentation of disease progression or death from any cause. Computed tomography/ magnetic resonance imaging (CT/MRI) scan at the conclusion of idelalisib monotherapy will serve as the reference for progression.
Pharmacokinetic Parameter: Cmax of Idelalisib | Predose and up to 24 hours postdose on Day 1 and Cycle 1, Day 5 of idelalisib + RICE combination therapy
  Cmax is defined as the maximum observed concentration of drug.
Pharmacokinetic Parameter: Cmax of GS-563117 | Predose and up to 24 hours postdose on Day 1 and Cycle 1, Day 5 of idelalisib + RICE combination therapy
  GS-563117 is the metabolite of idelalisib. Cmax is defined as the maximum observed concentration of drug.
Pharmacokinetic Parameter: Ctrough of Idelalisib | Predose and up to 24 hours postdose on Day 1 and Cycle 1, Day 5 of idelalisib + RICE combination therapy
  Ctrough is defined as the plasma concentration at the end of the dosing interval.
Pharmacokinetic Parameter: Ctrough of GS-563117 | Predose and up to 24 hours postdose on Day 1 and Cycle 1, Day 5 of idelalisib + RICE combination therapy
  Ctrough is defined as the plasma concentration at the end of the dosing interval.
Pharmacokinetic Parameter: Area Under the Concentration-Time Curve (AUC) of Idelalisib | Predose and up to 24 hours postdose on Day 1 and Cycle 1, Day 5 of idelalisib + RICE combination therapy
  AUC is defined as the plasma concentration at the end of the dosing interval.
Pharmacokinetic Parameter: Area Under the Concentration-Time Curve (AUC) of GS-563117 | Predose and up to 24 hours postdose on Day 1 and Cycle 1, Day 5 of idelalisib + RICE combination therapy
  AUC is defined as the plasma concentration at the end of the dosing interval.
Levels of Optional Exploratory Biomarkers on Bone Marrow Samples (eg pAKT, pS6 ribosomal protein) and plasma cytokines | Baseline and Day 21
Acceptability and Palatability of Idelalisib 10-mg Dispersible Tablet | Day 1 of idelalisib monotherapy and at Day 1, Cycle 1 of idelalisib in combination with RICE chemoimmunotherapy
  For participants who cannot swallow a whole tablet, the investigator will ask if the tablet administered as a suspension is palatable and will observe if the participant is able to swallow the dosage form. The acceptability and palatability of idelalisib dispersible tablets administered as an oral suspension (for participants unable to swallow the tablet) will be evaluated by a questionnaire administered to the participant and/or the parent/legal guardian.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- Centre Hospitalier Régional Universitaire de Lille, Lille, France
- Italy (3):
  - Istituto Giannina Gaslini, Genova
  - Ospedale Pediatrico Bambino Gesu, Roma
  - Infantile Regina Margherita Hospital, Torino
- Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw, Poland
- Spain (2):
  - Hospital Vall d´Hebrón, Barcelona
  - Hospital Universitario HM Monteprincipe, Madrid